CLINICAL TRIAL: NCT01429714
Title: Individually Tailored Elastic Compression Therapy After Deep Venous Thrombosis in Relation to the Incidence of Post Thrombotic Syndrome, a Randomized Multicenter Trial
Brief Title: The Ideal Deep Venous Thrombosis (DVT) Study
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-2-026; 80-82310-97-11017 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2011-08-24; First posted 2011-09-07 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Postthrombotic Syndrome
Keywords: Elastic Compression Stockings; Deep Venous Thrombosis; Post Thrombotic Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: individually tailored ECS (Experimental): Individually tailored duration of elastic compression therapy, based on signs and symptoms according to the Villalta scale, following an initial therapeutic period of 6 months.
  Interventions: Device: Individually tailored duration of elastic compression therapy
- Control: ECS 24 months (Active Comparator): Elastic compression therapy with a standard duration of 24 months
  Interventions: Device: Elastic compression therapy with a standard duration of 24 months

INTERVENTIONS:
Device: Individually tailored duration of elastic compression therapy — Individually tailored duration of elastic compression therapy,based on signs and symptoms according to the Villalta scale, following an initial therapeutic period of 6 months
  Other Names: Custom made flat knitted, knee length, class III stockings (Mediven ®550, ankle pressure 40 mmHg)
  Arms: Intervention: individually tailored ECS
Device: Elastic compression therapy with a standard duration of 24 months — Elastic compression therapy with a standard duration of 24 months
  Other Names: Custom made flat knitted, knee length, class III stockings (Mediven ®550, ankle pressure 40 mmHg)
  Arms: Control: ECS 24 months

SUMMARY:
In the Netherlands, 25.000 patients each year are diagnosed with Deep Venous Thrombosis (DVT). Elastic compression stocking (ECS) therapy reduces the incidence of post thrombotic syndrome (PTS) following DVT from 50% without ECS to 20-30% after ECS therapy for two years. It is however unclear whether all patients benefit to the same extent from this therapy or what the optimal duration of ECS therapy for individual patients should be. ECS therapy is not only costly, inconvenient and demanding but sometimes also even debilitating. Substantial costs could be saved by tailoring therapy to individual needs and as a result the quality of life for individual patients can be expected to improve.

This study aims to assess the costs and effects of tailoring the duration of ECS therapy after DVT to individual patients needs.

ECS therapy with a standard duration of 24 months will be compared with tailored ECS therapy, following an initial therapeutic period of 6 months, in patients with acute proximal DVT. The primary outcome is the percentage of patients with PTS at two year follow-up.

This is a multi-center, randomized, allocation concealed, single-blinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Legal age (18 yrs)
* Informed consent
* Acute objectively documented DVT of the leg
* Adequate anticoagulation

Exclusion Criteria:

* Previous DVT in the affected leg
* Recurrent DVT in the first 6 months following inclusion
* Preexistent venous insufficiency (skin signs C4-C6 on CEAP score or requiring ECS therapy)
* Contraindication for elastic compression therapy (arterial insufficiency)
* Active thrombolysis
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2011-03-22; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of PTS at 24 months after the event of acute DVT | At 24 months after the event of the acute DVT

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQOL) | Baseline, 3, 6, 12 and 24 months
  HRQOL, will be measured by questionnaires SF-36, EuroQol-5D, Veines-Qol Dutch translated
Recurrent venous thrombosis | 24 months
Mortality due to venous thrombosis | 24 months
Costs | 3, 6, 12, 24 months
  Costs will include direct costs (e.g. medical therapy) and indirect costs (e.g. travel) and will be measured by case record forms, hospital data and 5 retrospective cost-questionnaires
Patient Preferences | baseline, 24 months
  Patient preferences will be elicited by conducting a discrete choice experiment (DCE)

CONTACTS AND LOCATIONS:
Overall Officials: Arina J ten Cate-Hoek, MD, PhD, MpH, Principal Investigator — Maastricht University Medical Centre
Locations (14):
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua
  - Treviso Aziende, Treviso
- Netherlands (12):
  - Flevohospital, Almere Stad
  - VU Medical Centre, Amsterdam
  - Slotervaart hospital, Amsterdam
  - OLVG, Amsterdam
  - AMC, Amsterdam
  - Maxima Medical Centre, Eindhoven
  - UMCG, Groningen
  - Atrium Medical Centre, Heerlen
  - Westfriesgasthuis, Hoorn
  - Maastricht University Medical Centre, Maastricht
  - UMC Nijmegen Radboud, Nijmegen
  - Laurentius ziekenhuis, Roermond

REFERENCES:
- [Background] Ten Cate-Hoek AJ, Bouman AC, Joore MA, Prins M, Ten Cate H; IDEAL DVT trial investigators. The IDEAL DVT study, individualised duration elastic compression therapy against long-term duration of therapy for the prevention of post-thrombotic syndrome: protocol of a randomised controlled trial. BMJ Open. 2014 Sep 4;4(9):e005265. doi: 10.1136/bmjopen-2014-005265. PMID 25190617
- [Background] Ten Cate-Hoek AJ, Amin EE, Bouman AC, Meijer K, Tick LW, Middeldorp S, Mostard GJM, Ten Wolde M, van den Heiligenberg SM, van Wissen S, van de Poel MH, Villalta S, Serne EH, Otten HM, Klappe EH, Bistervels IM, Lauw MN, Piersma-Wichers M, Prandoni P, Joore MA, Prins MH, Ten Cate H; IDEAL DVT investigators. Individualised versus standard duration of elastic compression therapy for prevention of post-thrombotic syndrome (IDEAL DVT): a multicentre, randomised, single-blind, allocation-concealed, non-inferiority trial. Lancet Haematol. 2018 Jan;5(1):e25-e33. doi: 10.1016/S2352-3026(17)30227-2. Epub 2017 Dec 5. PMID 29217387
- [Derived] Iding AFJ, Ten Cate V, Ten Cate H, Wild PS, Ten Cate-Hoek AJ. Untangling profiles of postthrombotic syndrome using unsupervised machine learning. Blood Adv. 2025 Jul 22;9(14):3631-3641. doi: 10.1182/bloodadvances.2025015829. PMID 40086064
- [Derived] Amin EE, Ten Cate-Hoek AJ, Bouman AC, Meijer K, Tick L, Middeldorp S, Mostard G, Ten Wolde M, van den Heiligenberg S, van Wissen S, van de Poel M, Villalta S, Serne E, Otten HM, Klappe E, Prandoni P, Prins MH, Ten Cate H, Joore MA. Individually shortened duration versus standard duration of elastic compression therapy for prevention of post-thrombotic syndrome: a cost-effectiveness analysis. Lancet Haematol. 2018 Nov;5(11):e512-e519. doi: 10.1016/S2352-3026(18)30151-0. Epub 2018 Oct 9. PMID 30314712
- [Derived] Amin EE, Bistervels IM, Meijer K, Tick LW, Middeldorp S, Mostard G, van de Poel M, Serne EH, Otten HM, Klappe EM, Joore MA, Ten Cate H, Ten Wolde M, Ten Cate-Hoek AJ. Reduced incidence of vein occlusion and postthrombotic syndrome after immediate compression for deep vein thrombosis. Blood. 2018 Nov 22;132(21):2298-2304. doi: 10.1182/blood-2018-03-836783. Epub 2018 Sep 20. PMID 30237155
- [Derived] Amin EE, Joore MA, Ten Cate H, Meijer K, Tick LW, Middeldorp S, Mostard GJM, Ten Wolde M, van den Heiligenberg SM, van Wissen S, van de Poel MHW, Villalta S, Serne EH, Otten HM, Klappe EH, Prandoni P, Ten Cate-Hoek AJ. Clinical and economic impact of compression in the acute phase of deep vein thrombosis. J Thromb Haemost. 2018 Jun 1. doi: 10.1111/jth.14163. Online ahead of print. PMID 29856509